CLINICAL TRIAL: NCT00928278
Title: An Open Study To Estimate The Plasma Pharmacokinetics Of PF-04764793 Administered Via Oral Inhalation Using Dry Powder Inhalers.
Brief Title: A Study Estimating The Time Course Of PF-04764793 In The Blood Following Dosing By Oral Inhalation From Dry Powder Inhalers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B1691001; NCT00977535 (obsolete NCT alias)
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2009-12-21 (Estimated); Status verified 2009-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A - PF-04764793 (Experimental): PF-04764793 using inhaler A
  Interventions: Drug: Treatment A
- Treatment B - PF-04764793 (Active Comparator): PF-04764793 using inhaler B
  Interventions: Drug: Treatment B
- Treatment C - PF-04764793 (Experimental): PF-04764793 using inhaler A
  Interventions: Drug: Treatment C
- Treatment D - PF-04764793 (Active Comparator): PF-04764793 using inhaler B
  Interventions: Drug: Treatment D

INTERVENTIONS:
Drug: Treatment A — Inhaled, 300/150, single dose
  Arms: Treatment A - PF-04764793
Drug: Treatment B — Inhaled, 300/150, single dose
  Arms: Treatment B - PF-04764793
Drug: Treatment C — Inhaled, 300/150, single dose + oral activated charcoal block
  Arms: Treatment C - PF-04764793
Drug: Treatment D — Inhaled, 300/150, single dose + oral activated charcoal block
  Arms: Treatment D - PF-04764793

SUMMARY:
The purpose of this study is to investigate the time course of PF-04764793 concentration in the blood following dosing by oral inhalation from dry powder inhalers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 21 and 55 years.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m^2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males.
* Pregnant or nursing females.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic parameters: AUClast and Cmax | 48 hours

SECONDARY OUTCOMES:
Plasma pharmacokinetic parameters: AUC0-12, AUC0-24, AUCinf, Tmax and terminal half-life. | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1691001&StudyName=A%20Study%20Estimating%20The%20Time%20Course%20Of%20PF-04764793%20In%20The%20Blood%20Following%20Dosing%20By%20Oral%20Inhalation%20From%20Dry%20Powder%20Inhalers